CLINICAL TRIAL: NCT04997343
Title: Neurophysiological Estimates of Cortical Grey and White Matters Damage in Patients With Multiple Sclerosis
Brief Title: Neurophysiological Assessment in Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Antonella Conte, MD, Professor, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 6357
Record Dates: First submitted 2021-07-12; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Multiple Sclerosis; Demyelinating Disease; Inflammatory Disease
Keywords: neurophysiology; TMS-EEG; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases

STUDY DESIGN:
Intervention Model Description: In this multicenter, longitudinal, interventional (for TMS-EEG) -observational (for clinical and radiological variables obtained according to clinical practice) case-control study, all participants will undergo clinical and neurophysiological evaluation at baseline (T0). The baseline will consider the radiological data of disease activity. These evaluations will be repeated according to clinical practice in patients taking Disease modifying therapies (DMTs) or every 6 months, in a stable condition or according to the indication of the treating neurologist in case of disease reactivation. A one-year neurophysiological, clinical and radiological observation is foreseen. Healthy subjects will undergo only the neurophysiological evaluation at baseline. For the study, no hospital diagnostic equipment will be used, but machinery present in the research laboratories, for research use only, bearing the CE mark.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MS patients (Experimental): All MS patients will undergo clinical and neurophysiological evaluation at baseline (T0). The baseline will consider the radiological data of disease activity obtained from the most recently performed MRI according to clinical practice. These evaluations will be repeated according to clinical practice in patients taking DMT or every 6 months, in a stable condition or according to the indication of the treating neurologist in case of disease reactivation. A one-year neurophysiological, clinical and radiological observation is foreseen. Healthy subjects will undergo only the neurophysiological evaluation at baseline.
  Interventions: Other: Neurophysiological assessment; Other: clinical assessment
- Healthy controls (Other): Healthy subjects will undergo only the neurophysiological evaluation at baseline.
  Interventions: Other: Neurophysiological assessment

INTERVENTIONS:
Other: Neurophysiological assessment — EMG will be recorded from the Abductor pollicis brevis muscle (APB) with surface electrodes. EEG will be recorded with a 32-channel elastic cap via a TMS compatible system. TMS will be performed using a Magstim 200 stimulator with a 90 mm figure-of-eight coil localized on motor and non-motor areas using a neuronavigation system together with an optical tracking system. Coordinates for neuronavigation will be calculated in the MNI space and fit of each participant's anatomical MRI. Three minutes of continuous-EEG will be recorded with subjects at rest. Single-pulse neuronavigated TMS (sp-TMS) will be delivered at rest below the resting motor threshold intensity (RMT) over the APB hotspot on M1 during concurrent EEG recording. In a final block, the subject will maintain a voluntary muscle contraction (50% of the maximal voluntary contraction) of the left APB, and sp-TMS will be delivered at 130% RMT over the ipsilateral APB hotspot in order to record the lpSP.
Other: clinical assessment — Clinical evaluation, performed at each time point, will include:
  * The assessment of clinical disability using EDSS score
  * The multiple sclerosis functional composite (MSFC), a three-part quantitative objective measure of neurologic function, measuring lower limbs (timed 25-foot walk [T25FW]), upper limbs (nine-hole peg test [9HPT]) and cognitive (three-second paced auditory serial addition test [PASAT3]) function.
  In order to reduce inter-rater variability, the same physician/technician with adequate training will administer all three tests. The patient should feel comfortable with the situation. Examiner should explain the instructions in a professional but friendly way and let the patient ask any questions before starting the tests. Examiner should write down the test results, as well as any situation that disturbs the performance of patient. Examiner should not provide direct feedback to the patient about his/her performance
  Arms: MS patients

SUMMARY:
Main aim of this study will be the evaluation of the neurophysiological techniques of Transcranial Magnetic Stimulation (TMS) via electroencephalography (EEG) co-registration (TMS-EEG) with the study of TEPs (TEP: transcranial evoked potentials) as surrogates of white matter and grey matter functional integrity in patients with Multiple Sclerosis (MS). Data will be compared with those obtained from a group of healthy control subjects. Secondary aim will be the longitudinal evaluation of these neurophysiological parameters in MS patients during routine clinical and radiological evaluations, performed according to clinical practice, for 12 months.

To this aim a longitudinal multicenter study will be carried out, interventional (for neurophysiological techniques) and observational (for clinical and radiological evaluations), which involves the enrollment of 64 patients diagnosed with MS. Patients will keep their usual therapeutic regimen and their usual clinical-radiological checks according to clinical practice. The control group will consist of 64 healthy subjects, enrolled with prior written informed consent, age and sex-matched with MS patients and selected among the caregivers of the patients. Healthy subjects will only undergo neurophysiological assessment at baseline.

The neurophysiological evaluation will include the study of the propagation of potentials induced by stimulation. This method allows the study of cortical responses in terms of time domain and frequency, obtaining a measurement of interhemispheric connectivity and of microstructural and functional integrity of white matter. In the same way, these methods allow the assessment of grey matter integrity through the study of intracortical excitability.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a demyelinating disease of the central nervous system (CNS) whose pathogenesis involved both demyelinating events and neurodegeneration. It is on of the most frequent cause of disability in young adults. It is characterized by different clinical phenotypes: currently, the relapsing-remitting form (RR), the most common, and the progressive forms of MS (primary progressive -PP, secondary progressive -SP) are recognized. The relapsing-remitting form is characterized by the presence of acute/subacute onset of clinical events, the appearance of new lesions on magnetic resonance imaging (MRI), or the uptake of gadolinium by a new or pre-existing lesion. The progressive forms, on the other hand, present with a slow accumulation of disability from the onset (PP-MS), or following a relapsing-remitting trend (SP-MS). The clinical scale mainly used for evaluating patients with MS is the Expanded Disability Status Scale (EDSS). Currently, there are several treatments available for the control of the disease and the identification of the correct therapeutic choice can lead to an important slowdown, up to stabilization, of the clinical course of the disease. It is therefore essential, given the existence of different therapeutic strategies, to recognize early those patients who respond in a sub-optimal manner to therapy. To date, the evaluation of the effectiveness of the treatment is based on clinical and radiological data. Several studies have tried to identify new markers of disability, but none of these have entered the routine clinical use. In this context, the possible role of neurophysiology in early identify markers of inflammatory/ degenerative disease activity is outlined.

Among the neurophysiological methods potentially able to identify the inflammatory or neurodegenerative phase of the disease, the most promising results were obtained with transcranial magnetic stimulation (TMS) and electroencephalography (EEG). These methods, already widely used in the clinical setting, are characterized by being reproducible, non-invasive and low-cost. Thanks to the development of EEG systems compatible with magnetic stimulation, it is possible to study the cortical potentials evoked by TMS (TEPs). The TEPs constitute a sensitive and reproducible experimental index of intracortical excitability and allow the identification of specific alterations of different neurological conditions. The study of TEPs offers a better performance than that obtainable using the single techniques, TMS and EEG, separately.

Neurophysiological estimates of white matter integrity Several evidence have confirmed that the EEG indices of functional connectivity are influenced by the degree of myelination of the white matter. Among these indices of EEG connectivity, cortico-cortical coherence is a linear correlation index between the oscillatory signal of two cortical areas and has been shown to be a sensitive index of the myelination state of the brain in physiological conditions and in various neurological pathologies.

Distinct EEG oscillations in the different frequency bands revealed many robust relationships to behavioral, cognitive, and clinical states in several studies. Spatial-temporal oscillatory dynamic patterns recorded by EEG are important brain state-dependent measures of neocortical dynamics, including functional connectivity. Myelin is critical for sustaining oscillatory neural activity and entrainment between "generators" (e.g., cell assemblies or networks at multiple scales) in brain regions separated by substantial conduction delays. Functional connectivity as assessed by scalp EEG at large scales is believed to be strongly influenced by white matter tracts, especially the cortico-cortical projections. The standard Fourier transform-based multi-channel signal measure coherence is a squared correlation coefficient expressed as a function of frequency; it can provide robust measures of cognitive state and white matter (WM) maturation or disease. WM integrity determines propagation delays (i.e. the timing) of synaptic inputs in a determined brain network thus allowing phase synchrony of local oscillations. Relatively small changes in conduction delays can have significant effects on oscillatory coupling and phase synchrony between distant brain regions. Disruption in brain synchronization contributes to dysfunction in many neurological and psychiatric disorders. Compared to scalp EEG, high-resolution EEG (HR-EEG) methods employ computer algorithms (e.g., Laplacian or dura image) to provide estimates of brain or dural surface potentials at roughly the 2-3 cm scale. HR-EEG functional connectivity measures, like narrow band (e.g., 1 Hz) alpha and theta coherence, has been linked to cortico-cortical signal propagation via (mostly) myelinated axons. The propagation time between hemispheres is about 30 ms through myelinated callosal fibers and 150-300ms through unmyelinated fibers. An investigation of scalp-registered inter-hemispheric coherence between the left and right sensorimotor hand areas using HR-EEG revealed a superposition of both bilaterally coherent and incoherent rhythmic activities within the alpha band. Synaptic integration can be expected to be strongly influenced by the degree of myelination of intercallosal axons. Combined EEG and HR-EEG can provide complementary functional connectivity estimates that are maximally sensitive to large/global (~5-10 cm) and intermediate/local {-2-3 cm) spatial scale source regions, respectively. White matter integrity is important for cortico-cortical connections and is critical to these functional connectivity estimates, especially scalp oscillatory coupling and distant sources phase coherence.

Transcranial magnetic stimulation (TMS) is a non-invasive brain-stimulation technique. By producing high-intensity magnetic pulse, TMS induces brief electric currents that can excite or inhibit a small area of the cerebral cortex. This activating property is classically used on the primary motor cortex (M1) to produce action potentials along the cortico-spinal bundle and evoke a motor potential (MEP, motor evoked potential) in the contralateral musculature. In MS patients, EEG and TMS are widely used as diagnostic tools to prove demyelination by means of abnormal conduction time along white matter tracts, even in subjects with normal MRI scans. Furthermore, when the magnetic stimulus is delivered during voluntary muscle contraction of the stimulation target muscle, the TMS of M1 can generate a brief interruption of voluntary electromyography (EMG) activity both contralateral (CSP: contralateral silent period) and ipsilateral (the " ipsilateral silent period" -IpSP). lpSP is a measure of interhemispheric motor inhibition that has been found to be altered in patient with MS and callosal lesions.

Compared to the separate recording of the EEG signals and those generated by the TMS, the simultaneous execution of the two methods - TMS-EEG - allows the recording directly from the scalp of the potentials (TEP) evoked by the TMS. The recording of TEPs from areas distant from the stimulation site allows to obtain information about the connectivity of the stimulated cortex. The "interhemispheric signal propagation" (ISP) is a measure of interhemispheric connectivity based on the propagation of TMS-EEG responses from the stimulated hemisphere to the contralateral. The ISP correlates with the microstructural integrity of the callosal microfibers and with the hand dexterity during motor development.

Neurophysiological estimates of grey matter Integrity:

Regarding gray matter (GM) pathology, evidences obtained from TMS and EEG studies have contributed to unveil the role of cortical dysfunction in MS. Alterations in EEG oscillations considered important in sensorimotor integration and motor control have been associated with clinical disorders and radiological changes in patients with MS. Furthermore, paired-pulse TMS protocols have shown alterations in M1 excitability in MS patients and that these alterations correlate with clinical disability. Among the measures of TMS-EEG, the locally recorded TEPs reflect the excitability and activation state of the stimulated cortex and therefore the degree of integrity of the cortical gray matter.

In conclusion, EEG and TMS-EEG measures are powerful tools to assess WM and GM functional integrity in patients with MS. As such, EEG and TMS-EEG also provide a potential objective framework to systematically assess the efficacy of Disease modifying therapies (DMTs) in MS.

Study aims and hypotheses Main aim of this study is the evaluation of TMS-EEG neurophysiological measures as surrogates of functional integrity of both gray and white matter in MS patients. The data obtained will be compared with those of a group of healthy subjects comparable for sex and age. Healthy subjects will be identified as those with normal neurological examination and negative medical history for morbidity. By combining the neurophysiological variables with the clinical ones, an attempt will be made to identify neurophysiological markers expressing the degree of disability of patients with MS (primary objective). The secondary objective is to identify the neurophysiological variables that may play a predictive role in the clinical or radiological relapses of the pathology and of the long-term clinical-radiological status. To this aim, the neurophysiological TMS-EEG measurements will be repeated longitudinally in the patients participating in the study and correlated with the clinical and radiological according to clinical practice. The neurophysiological markers identified may offer support in identifying patients in clinical deterioration or with a sub-optimal response to therapy.

Enrollment: To guarantee an adequate number of study participants and obtain data that are more traceable to real-life conditions, the investigators will collaborate in recruiting with other MS Centers (list with the relevant Managers attached). All neurophysiological evaluations will be performed at our Department and our Center will be the coordinator.

Tolerability of the neurophysiological evaluation The selected neurophysiological methods are non-invasive procedures, widely used and based on tools currently in use in clinical practice. These methods are painless and therefore easily implemented in a large population of subjects as they are safe and free of side effects.

ELIGIBILITY:
Inclusion Criteria:

* MS diagnosis according to the latest McDonald criteria

Exclusion Criteria:

* other neurological or immunological diseases
* clinical relapses in the 30 days prior to the clinical and neurophysiological evaluation;
* presence of conditions that contraindicate the execution of Transcranial Magnetic Stimulation (TMS) methods (history of epilepsy, pacemaker, recent head injury).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Global cortico-cortical myelination | Baseline (T0) and at 6 and 12 months. Healthy controls will undergo only the neurophysiological evaluation at baseline.
  Power of the dominant frequency peak of the global electroencephalography (EEG) signal.
Changes of the Cortical-cortical coherence | Baseline (T0) and at 6 and 12 months. Healthy controls will undergo only the neurophysiological evaluation at baseline.
  Coherence between EEG signals recorded from distant channels.
Changes of the Local cortical-cortical myelination (motor) | Baseline (T0) and at 6 and 12 months. Healthy controls will undergo only the neurophysiological evaluation at baseline.
  Power of the dominant frequency peak of the local EEG signal on primary motor cortex (M1).
Changes of the Trans-callosal axonal myelination | Baseline (T0) and at 6 and 12 months. Healthy controls will undergo only the neurophysiological evaluation at baseline.
  Cortico-cortical coherence between EEG signals recorded on primary motor cortex (M1) areas bilaterally.
Changes of Interhemispheric signal propagation (iSP) | Baseline (T0) and at 6 and 12 months. Healthy controls will undergo only the neurophysiological evaluation at baseline.
  TMS-EMG measurement of the ipsilateral silent period (IpSP)
Changes of TMS-EEG measurement of the functional integrity of the grey matter: | Baseline (T0) and at 6 and 12 months. Healthy controls will undergo only the neurophysiological evaluation at baseline.
  Amplitude of the early components of Transcranial evoked potentials (TEPs).
Changes of TMS-EMG measurement of the functional integrity of the grey matter: | Baseline (T0) and at 6 and 12 months. Healthy controls will undergo only the neurophysiological evaluation at baseline.
  Resting Motor Threshold- (RMT)
Changes of clinical outcome measures | Baseline (T0) and at 6 and 12 months. Healthy controls will undergo only the neurophysiological evaluation at baseline.
  Clinical disability will be monitored with the Expanded Disability Status Scale (EDSS), performed by the same neurologist at each timepoint.
Changes of the Multiple Sclerosis Functional Composite (MSFC) | Baseline (T0) and at 6 and 12 months. Healthy controls will undergo only the neurophysiological evaluation at baseline.
  To assess walking, lower limb functionality, upper limb dexterity and cognitive function.
Changes of radiological outcome measures | Baseline (T0) and at 6 and 12 months. Healthy controls will undergo only the neurophysiological evaluation at baseline.
  Evaluation of the lesion load
Changes of magnetic resonance imaging (MRI) number of lesions in T2 | Baseline (T0) and at 6 and 12 months. Healthy controls will undergo only the neurophysiological evaluation at baseline.
  Evaluation of new lesions in T2 compared to the previous evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Centonze, MD, PhD, Principal Investigator — Unit of Neurology, IRCCS Neuromed, Pozzilli, IS

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD will be shared at the end of the study by request from any qualified investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 3 months after data pubblication
Access Criteria: research group focused in neurophysiological investigations in patients with multiple sclerosis

REFERENCES:
- [Background] Boniface SJ, Mills KR, Schubert M. Responses of single spinal motoneurons to magnetic brain stimulation in healthy subjects and patients with multiple sclerosis. Brain. 1991 Feb;114 ( Pt 1B):643-62. doi: 10.1093/brain/114.1.643. PMID 2004261
- [Background] Casula EP, Maiella M, Pellicciari MC, Porrazzini F, D'Acunto A, Rocchi L, Koch G. Novel TMS-EEG indexes to investigate interhemispheric dynamics in humans. Clin Neurophysiol. 2020 Jan;131(1):70-77. doi: 10.1016/j.clinph.2019.09.013. Epub 2019 Oct 24. PMID 31756594
- [Background] Conte A, Lenzi D, Frasca V, Gilio F, Giacomelli E, Gabriele M, Bettolo CM, Iacovelli E, Pantano P, Pozzilli C, Inghilleri M. Intracortical excitability in patients with relapsing-remitting and secondary progressive multiple sclerosis. J Neurol. 2009 Jun;256(6):933-8. doi: 10.1007/s00415-009-5047-0. Epub 2009 Mar 1. PMID 19252788
- [Background] Cutter GR, Baier ML, Rudick RA, Cookfair DL, Fischer JS, Petkau J, Syndulko K, Weinshenker BG, Antel JP, Confavreux C, Ellison GW, Lublin F, Miller AE, Rao SM, Reingold S, Thompson A, Willoughby E. Development of a multiple sclerosis functional composite as a clinical trial outcome measure. Brain. 1999 May;122 ( Pt 5):871-82. doi: 10.1093/brain/122.5.871. PMID 10355672
- [Background] Dobson R, Giovannoni G. Multiple sclerosis - a review. Eur J Neurol. 2019 Jan;26(1):27-40. doi: 10.1111/ene.13819. Epub 2018 Nov 18. PMID 30300457
- [Background] Ferrazzano G, Crisafulli SG, Baione V, Tartaglia M, Cortese A, Frontoni M, Altieri M, Pauri F, Millefiorini E, Conte A. Early diagnosis of secondary progressive multiple sclerosis: focus on fluid and neurophysiological biomarkers. J Neurol. 2021 Oct;268(10):3626-3645. doi: 10.1007/s00415-020-09964-4. Epub 2020 Jun 5. PMID 32504180
- [Background] Giovannoni G, Lang S, Wolff R, Duffy S, Hyde R, Kinter E, Wakeford C, Sormani MP, Kleijnen J. A Systematic Review and Mixed Treatment Comparison of Pharmaceutical Interventions for Multiple Sclerosis. Neurol Ther. 2020 Dec;9(2):359-374. doi: 10.1007/s40120-020-00212-5. Epub 2020 Sep 28. PMID 32989721
- [Background] Goodkin DE, Hertsgaard D, Seminary J. Upper extremity function in multiple sclerosis: improving assessment sensitivity with box-and-block and nine-hole peg tests. Arch Phys Med Rehabil. 1988 Oct;69(10):850-4. PMID 3178453
- [Background] Hallett M. Transcranial magnetic stimulation: a primer. Neuron. 2007 Jul 19;55(2):187-99. doi: 10.1016/j.neuron.2007.06.026. PMID 17640522
- [Background] Houdayer E, Comi G, Leocani L. The Neurophysiologist Perspective into MS Plasticity. Front Neurol. 2015 Sep 3;6:193. doi: 10.3389/fneur.2015.00193. eCollection 2015. PMID 26388835
- [Background] Jarczok TA, Fritsch M, Kroger A, Schneider AL, Althen H, Siniatchkin M, Freitag CM, Bender S. Maturation of interhemispheric signal propagation in autism spectrum disorder and typically developing controls: a TMS-EEG study. J Neural Transm (Vienna). 2016 Aug;123(8):925-35. doi: 10.1007/s00702-016-1550-5. Epub 2016 May 13. PMID 27177879
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Lenzi D, Conte A, Mainero C, Frasca V, Fubelli F, Totaro P, Caramia F, Inghilleri M, Pozzilli C, Pantano P. Effect of corpus callosum damage on ipsilateral motor activation in patients with multiple sclerosis: a functional and anatomical study. Hum Brain Mapp. 2007 Jul;28(7):636-44. doi: 10.1002/hbm.20305. PMID 17080438
- [Background] Leocani L, Colombo B, Magnani G, Martinelli-Boneschi F, Cursi M, Rossi P, Martinelli V, Comi G. Fatigue in multiple sclerosis is associated with abnormal cortical activation to voluntary movement--EEG evidence. Neuroimage. 2001 Jun;13(6 Pt 1):1186-92. doi: 10.1006/nimg.2001.0759. PMID 11352624
- [Background] Leocani L, Rovaris M, Martinelli-Boneschi F, Annovazzi P, Filippi M, Colombo B, Martinelli V, Comi G. Movement preparation is affected by tissue damage in multiple sclerosis: evidence from EEG event-related desynchronization. Clin Neurophysiol. 2005 Jul;116(7):1515-9. doi: 10.1016/j.clinph.2005.02.026. Epub 2005 Apr 26. PMID 15953556
- [Background] Lublin FD, Reingold SC, Cohen JA, Cutter GR, Sorensen PS, Thompson AJ, Wolinsky JS, Balcer LJ, Banwell B, Barkhof F, Bebo B Jr, Calabresi PA, Clanet M, Comi G, Fox RJ, Freedman MS, Goodman AD, Inglese M, Kappos L, Kieseier BC, Lincoln JA, Lubetzki C, Miller AE, Montalban X, O'Connor PW, Petkau J, Pozzilli C, Rudick RA, Sormani MP, Stuve O, Waubant E, Polman CH. Defining the clinical course of multiple sclerosis: the 2013 revisions. Neurology. 2014 Jul 15;83(3):278-86. doi: 10.1212/WNL.0000000000000560. Epub 2014 May 28. PMID 24871874
- [Background] Mori F, Kusayanagi H, Monteleone F, Moscatelli A, Nicoletti CG, Bernardi G, Centonze D. Short interval intracortical facilitation correlates with the degree of disability in multiple sclerosis. Brain Stimul. 2013 Jan;6(1):67-71. doi: 10.1016/j.brs.2012.02.001. Epub 2012 Feb 24. PMID 22425067
- [Background] Murias M, Webb SJ, Greenson J, Dawson G. Resting state cortical connectivity reflected in EEG coherence in individuals with autism. Biol Psychiatry. 2007 Aug 1;62(3):270-3. doi: 10.1016/j.biopsych.2006.11.012. Epub 2007 Mar 6. PMID 17336944
- [Background] Noseworthy JH, Lucchinetti C, Rodriguez M, Weinshenker BG. Multiple sclerosis. N Engl J Med. 2000 Sep 28;343(13):938-52. doi: 10.1056/NEJM200009283431307. No abstract available. PMID 11006371
- [Background] Nunez PL, Srinivasan R. A theoretical basis for standing and traveling brain waves measured with human EEG with implications for an integrated consciousness. Clin Neurophysiol. 2006 Nov;117(11):2424-35. doi: 10.1016/j.clinph.2006.06.754. Epub 2006 Sep 22. PMID 16996303
- [Background] Nunez PL, Westdorp AF. The surface Laplacian, high resolution EEG and controversies. Brain Topogr. 1994 Spring;6(3):221-6. doi: 10.1007/BF01187712. PMID 8204409
- [Background] Pajevic S, Basser PJ, Fields RD. Role of myelin plasticity in oscillations and synchrony of neuronal activity. Neuroscience. 2014 Sep 12;276:135-47. doi: 10.1016/j.neuroscience.2013.11.007. Epub 2013 Nov 28. PMID 24291730
- [Background] Srinivasan R. Spatial structure of the human alpha rhythm: global correlation in adults and local correlation in children. Clin Neurophysiol. 1999 Aug;110(8):1351-62. doi: 10.1016/s1388-2457(99)00080-2. PMID 10454270
- [Background] Thatcher RW, Krause PJ, Hrybyk M. Cortico-cortical associations and EEG coherence: a two-compartmental model. Electroencephalogr Clin Neurophysiol. 1986 Aug;64(2):123-43. doi: 10.1016/0013-4694(86)90107-0. PMID 2424729
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Tremblay S, Rogasch NC, Premoli I, Blumberger DM, Casarotto S, Chen R, Di Lazzaro V, Farzan F, Ferrarelli F, Fitzgerald PB, Hui J, Ilmoniemi RJ, Kimiskidis VK, Kugiumtzis D, Lioumis P, Pascual-Leone A, Pellicciari MC, Rajji T, Thut G, Zomorrodi R, Ziemann U, Daskalakis ZJ. Clinical utility and prospective of TMS-EEG. Clin Neurophysiol. 2019 May;130(5):802-844. doi: 10.1016/j.clinph.2019.01.001. Epub 2019 Jan 19. PMID 30772238
- [Background] Voineskos AN, Farzan F, Barr MS, Lobaugh NJ, Mulsant BH, Chen R, Fitzgerald PB, Daskalakis ZJ. The role of the corpus callosum in transcranial magnetic stimulation induced interhemispheric signal propagation. Biol Psychiatry. 2010 Nov 1;68(9):825-31. doi: 10.1016/j.biopsych.2010.06.021. Epub 2010 Aug 12. PMID 20708172